CLINICAL TRIAL: NCT00193791
Title: Concomitant Chemo-radiation in Advanced Stage Carcinoma Cervix: A Phase III Randomized Trial
Brief Title: Concomitant Chemoradiation in Advanced Stage Carcinoma Cervix
Acronym: CRACx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Sk Shrivastava, Professor and Head, Radiation Oncology, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH/114/2003/CRACX TRIAL
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Cancer of Cervix
Keywords: Carcinoma Cervix; FIGO Stage IIIB; Radiation therapy; Chemoradiation; Treatment related toxicities; Cervical Cancer; Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Concomitant chemo-radiation versus radiation alone
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation (RT) Alone (No Intervention): Standard radical radiation therapy alone
- CT + RT (Experimental): Injection Cisplatin 40mg/m2 weekly for 5 weeks during the entire course of external radiation therapy
  Interventions: Other: CT + RT

INTERVENTIONS:
Other: CT + RT — Injection Cisplatin 40mg/m2 weekly for 5 weeks during the entire course of external radiation therapy
  Arms: CT + RT

SUMMARY:
A study to evaluate the efficacy of concomitant chemoradiation as compared to radiotherapy alone. Concomitant chemoradiation is not a new treatment modality for carcinoma cervix. Studies have shown improvement in survivals with chemoradiation, but majority of the patients was in early stages. Since this treatment modality has not been tested adequately in advanced stages in our setting, the present study is being undertaken. The study arm of chemoradiation has the potential to improve the survivals by 10%, but is associated with additional 5% risk of toxicities, which are treatable. In the study arm, apart form the standard radiotherapy treatment, you will receive weekly chemotherapy injections (Cisplatin) during external radiation therapy. The study arm is associated with additional 5% acute hematological and gastrointestinal toxicities, which are treatable with medications, blood transfusions, modifications in the ongoing treatment etc.

DETAILED DESCRIPTION:
Carcinoma cervix is the commonest malignancy seen in Asian women and constitutes approximately 30% of all cancers (1). It is also the leading cause of cancer mortality in India. Nearly 50% of the patients present with advanced stages (FIGO Stage III/IV). The main stay of treatment has traditionally been radical radiation therapy and over decades the survival rates have achieved a plateau of 30 - 45% at 5 years. In developing countries the socioeconomic problems, illiteracy, late presentation and irregular follow-up have further compromised our survivals. Over the last decade there have been studies on the use of chemo-radiotherapy in carcinoma cervix. Over 19 randomized trials have been published addressing the issue of chemo-radiotherapy. However, heterogeneous data, poor randomization, inadequate number of patients, sub-optimal radiotherapy, non-uniform use of chemotherapeutic drugs, its sequencing and poor documentation have not yet provided the evidence to substantially alter the practice. Hence, meta-analysis of these trials was undertaken to further evaluate the role of chemo-radiotherapy in carcinoma cervix (2,3).

The first meta-analysis published by Cochrane Collaborative Group of 4580 randomized patients (19 randomized trials) suggested that chemo-radiation did show an absolute survival benefit improvement both in progression free and overall survivals by 16% and 12% respectively (p<0.0001). The survivals were significantly better with Cisplatin based concomitant chemo-radiation (p<0.0001). Incidentally, the distant metastasis rates were also significantly lower in chemo-radiation (p<0.0001). However, all these benefits were seen only in early stages. In addition, acute grade 3/4 hematological and gastro-intestinal toxicities were higher with chemo-radiation (additional 8% and 5% respectively). The data was insufficient to report on late toxicity (2).

The second meta-analysis of 9 randomized trials, recently published by the Canadian Group to evaluate only cisplatin based concomitant chemo-radiation confirms the improvement in overall survival (4year survival data) in advanced stages, bulky IB tumors (prior to surgery) and high risk early disease (post-surgery). Although acute grade 3/4 hematological and gastro-intestinal toxicities were higher in chemo-radiation, they were short-lived, with only 2 deaths and the remaining resolved with medical treatment. There was no significant increase in the late toxicity from the data available.

Both the Cochrane and Canadian meta-analysis have to a large extent tried to address the role of concomitant chemo-radiation, but Carcinoma Cervix Stage III accounted for only 30-35% and moreover evaluation with optimal radiation schedules and comparison of late toxicities still remains unanswered. What is more important is that the cisplatin is relatively inexpensive and is available worldwide. This means that cisplatin-based chemo-radiation is affordable in the developing countries where carcinoma cervix still forms the major cancer. However, the role of chemo-radiation in Carcinoma Cervix Stage IIIB in a developing countries including India still remains unexplored. We propose this randomized study to evaluate the role and benefit of chemo-radiation in-patients with cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous carcinoma of cervix
* Performance index world health organization (WHO) grade 0 or 1
* Patients below 65 years of age
* FIGO Stage IIIB
* Normal ECG and Cardiovascular system
* Normal hematological parameters
* Normal renal and liver function tests

Exclusion Criteria:

* Co-morbid conditions like medical renal disease
* Medical or Psychological condition that would preclude treatment
* H/o Previous treatment / Pregnancy
* Patient unreliable for treatment completion and follow-up.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2003-07-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To compare the disease free survivals. | December 2009

SECONDARY OUTCOMES:
To compare the overall survivals | December 2010
To compare the distant metastasis rates | December 2010
To compare the quality of life in both the groups | December 2010
To compare the normal tissue toxicities (Acute & Late) of standard radiation therapy with concomitant chemo-radiation. | June 2017

CONTACTS AND LOCATIONS:
Overall Officials: Shyamkishore J Shrivastava, MD,DNB(RT), Principal Investigator — Professor & Head, Department of Radiation Oncology, Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) related to patient characteristics, treatment and outcome variables.

REFERENCES:
- [Background] Green JA, Kirwan JM, Tierney JF, Symonds P, Fresco L, Collingwood M, Williams CJ. Survival and recurrence after concomitant chemotherapy and radiotherapy for cancer of the uterine cervix: a systematic review and meta-analysis. Lancet. 2001 Sep 8;358(9284):781-6. doi: 10.1016/S0140-6736(01)05965-7. PMID 11564482
- [Background] Lukka H, Hirte H, Fyles A, Thomas G, Elit L, Johnston M, Fung MF, Browman G; Cancer Care Ontario Practice Guidelines Initiative Gynecology Disease Site Group. Concurrent cisplatin-based chemotherapy plus radiotherapy for cervical cancer--a meta-analysis. Clin Oncol (R Coll Radiol). 2002 Jun;14(3):203-12. doi: 10.1053/clon.2002.0076. PMID 12109823
- [Derived] Shrivastava S, Mahantshetty U, Engineer R, Chopra S, Hawaldar R, Hande V, Kerkar RA, Maheshwari A, Shylasree TS, Ghosh J, Bajpai J, Gurram L, Gulia S, Gupta S; Gynecologic Disease Management Group. Cisplatin Chemoradiotherapy vs Radiotherapy in FIGO Stage IIIB Squamous Cell Carcinoma of the Uterine Cervix: A Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):506-513. doi: 10.1001/jamaoncol.2017.5179. PMID 29423520